CLINICAL TRIAL: NCT03859258
Title: A Prospective Controlled Ultrasound Based Study For Niche Development In The Uterine Cesarean Section Scar With Hysteroscopic Correlation In Symptomatizing Patients
Brief Title: Ultrasound Based Study For Niche Development In The Uterine Cesarean Section Scar
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Raafat Abdelfatah Mohamed Said, Assistant lecturer of obstetrics and gynecology, Cairo University
Other Study IDs: CSD1
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Cesarean Section; Dehiscence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient having Cesarean section: Transvaginal sonography for patients having ceserean section to assess uterine Niche development and parameters
  Interventions: Device: Transvaginal sonography
- Patient delivered vaginally: Transvaginal sonography for patients having vaginal delivery to confirm absence of uterine Niche development
  Interventions: Device: Transvaginal sonography

INTERVENTIONS:
Device: Transvaginal sonography — Niche is assessed using TVS, SIS (cases only) and office hysteroscopy
  Other Names: SIS, office hysteroscopy

SUMMARY:
The aim of this study is to evaluate different factors affecting niche development in the uterine cesarean section scar in women enrolled 3 to 6 months after cesarean delivery using both TVS and SIS.

DETAILED DESCRIPTION:
Cesarean delivery is amongst the most widely recognized operations performed on women and its rate continue expanding. The rates of cesarean section (CS) in the United States in 1996 and 2009 were 20.7% and 32.3% respectively, witnessing an expansion of more than half. In China, 50% of deliveries in 2010 were through CS. In the Netherlands, the cesarean delivery rate jumped from 7.4 to 15.8% between 1990 and 2008, whereas in the United Kingdom, the CS rate increased from 12 to 29% throughout the same time period. In Brazil, the CS rate jumped from 15% in 1970 to even 80% in 2004.

The expanding rate of cesarean deliveries can be credited to many variables including an increase in repeated cesarean sections. There is no discourse that CS is a lifesaving method for a few women, for instance for women with placenta previa or obstructed labor, or for fetuses with either antenatal or intrapartum distress, breech pregnancy or a twin pregnancy. The World Health Organization suggests that the ideal CS rate should be 15%.

Also, this expanding CS rate has fortified an enthusiasm for the potential long-term morbidity of CS scars. By and large, the cesarean incision heals uneventfully. However, some authors depicted a cesarean scar defect on transvaginal sonography (TVS) or saline infusion sonography (SIS) as a wedge shape anechoic structure at the site of the scar or a gap in anterior myometrium of the anterior lower myometrium at the site of previous cesarean section site. This was first described using hysterosalpingography in 1961. The terminology used to describe these scar abnormalities include scar defects, or 'niches' in the uterine scar, cesarean scar defect, uterine diverticulum, uterine isthmocele, pouch or sacculation and differs various publications. The term 'niche', which was introduced in 2001. A niche appears to be frequently present after a CS. Using SIS, niches were identified in the scar in more than half of the women who had had a caesarean delivery. Niches were defined as indentations of the myometrium of at least 2 mm. Large niches occur less frequently, with an incidence varying from 11 to 45% dependent on the definition used (a depth of at least 50 or 80% of the anterior myometrium, or the remaining myometrial thickness ≤2.2 mm when evaluated by TVS and ≤2.5 mm when evaluated by sonohysterography).

It is usually asymptomatic. Be that as it may, some authors have described some symptoms identified with this condition and there are several studies relating abnormal uterine bleeding and niche, especially postmenstrual spotting which appears to be the most common symptom in women with niches due to the collection of menstrual blood in a uterine scar defect causing postmenstrual spotting.

Later prospective cohort studies reported spotting in ∼30% of women with a niche at 6- 12 months after their CS compared with 15% of women without a niche after CS. It is undoubtedly a generally new pathology that needs assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Cases are delivered by Lower segment cesarean section
2. Controls are delivered vaginally
3. Singleton fetus
4. Living fetus
5. Term pregnancy

Exclusion Criteria:

1. Placenta praevia
2. Congenital fetal anomalies
3. Severe oligohydramnios(MVP <2cm)
4. Rupture of membranes more than 18 hours
5. Puerperal pyrexia or sepsis
6. Bladder injury
7. Blood transfusion

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Rate of Niche development in the uterine cesarean section scar | baseline
  Measure number of patients that will develop uterine Niche following lower segment cesarean section

SECONDARY OUTCOMES:
Measuring Residual myometrial thickness (RMT) | baseline
  Measuring the remaining myometrium above uterine Niche
Measuring depth of uterine Niche | baseline
  Measuring the depth of cesarean scar defect developed after cesarean section
Measuring width of uterine Niche | baseline
  Measuring the width of cesarean scar defect developed after cesarean section
Assessment of potential risk factors for Niche development | baseline
  Detect why Niche develop
Rate of postmenstrual spotting in patients with uterine Niche | baseline
  Measure number of patients having uterine Niche that will complain from postmenstrual spotting
Rate of uterine Isthmocele development on hysteroscopic evaluation in patients presenting with postmenstrual spotting after cesarean section | basline
  Measure number of patients having uterine Isthmocele detected during hysteroscopic evaluation from all patients presenting with postmenstrual spotting

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Aboulghar, M.D., Principal Investigator — Cairo University; Hassan M Gaafar, M.D., Principal Investigator — Cairo University; Hisham M Haggag, M.D., Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Barros AJ, Santos IS, Matijasevich A, Domingues MR, Silveira M, Barros FC, Victora CG. Patterns of deliveries in a Brazilian birth cohort: almost universal cesarean sections for the better-off. Rev Saude Publica. 2011 Aug;45(4):635-43. doi: 10.1590/s0034-89102011005000039. Epub 2011 Jun 10. PMID 21670862
- [Background] Betran AP, Merialdi M, Lauer JA, Bing-Shun W, Thomas J, Van Look P, Wagner M. Rates of caesarean section: analysis of global, regional and national estimates. Paediatr Perinat Epidemiol. 2007 Mar;21(2):98-113. doi: 10.1111/j.1365-3016.2007.00786.x. PMID 17302638
- [Background] Bij de Vaate AJ, Brolmann HA, van der Voet LF, van der Slikke JW, Veersema S, Huirne JA. Ultrasound evaluation of the Cesarean scar: relation between a niche and postmenstrual spotting. Ultrasound Obstet Gynecol. 2011 Jan;37(1):93-9. doi: 10.1002/uog.8864. PMID 21031351
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650
- [Background] Clark EA, Silver RM. Long-term maternal morbidity associated with repeat cesarean delivery. Am J Obstet Gynecol. 2011 Dec;205(6 Suppl):S2-10. doi: 10.1016/j.ajog.2011.09.028. Epub 2011 Oct 6. PMID 22114995
- [Background] Deng W, Klemetti R, Long Q, Wu Z, Duan C, Zhang WH, Ronsmans C, Zhang Y, Hemminki E. Cesarean section in Shanghai: women's or healthcare provider's preferences? BMC Pregnancy Childbirth. 2014 Aug 22;14:285. doi: 10.1186/1471-2393-14-285. PMID 25148697
- [Background] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016
- [Background] Feng XL, Wang Y, An L, Ronsmans C. Cesarean section in the People's Republic of China: current perspectives. Int J Womens Health. 2014 Jan 9;6:59-74. doi: 10.2147/IJWH.S41410. eCollection 2014. PMID 24470775
- [Background] Hofmeyr GJ, Hannah M, Lawrie TA. Planned caesarean section for term breech delivery. Cochrane Database Syst Rev. 2015 Jul 21;2015(7):CD000166. doi: 10.1002/14651858.CD000166.pub2. PMID 26196961
- [Background] Monteagudo A, Carreno C, Timor-Tritsch IE. Saline infusion sonohysterography in nonpregnant women with previous cesarean delivery: the "niche" in the scar. J Ultrasound Med. 2001 Oct;20(10):1105-15. doi: 10.7863/jum.2001.20.10.1105. PMID 11587017
- [Background] Naji O, Abdallah Y, Bij De Vaate AJ, Smith A, Pexsters A, Stalder C, McIndoe A, Ghaem-Maghami S, Lees C, Brolmann HA, Huirne JA, Timmerman D, Bourne T. Standardized approach for imaging and measuring Cesarean section scars using ultrasonography. Ultrasound Obstet Gynecol. 2012 Mar;39(3):252-9. doi: 10.1002/uog.10077. PMID 21858885
- [Background] Osser OV, Jokubkiene L, Valentin L. High prevalence of defects in Cesarean section scars at transvaginal ultrasound examination. Ultrasound Obstet Gynecol. 2009 Jul;34(1):90-7. doi: 10.1002/uog.6395. PMID 19499514
- [Background] Osterman MJ, Martin JA. Primary cesarean delivery rates, by state: results from the revised birth certificate, 2006-2012. Natl Vital Stat Rep. 2014 Jan;63(1):1-11. PMID 24461076
- [Background] POIDEVIN LO. The value of hysterography in the prediction of cesarean section wound defects. Am J Obstet Gynecol. 1961 Jan;81:67-71. doi: 10.1016/s0002-9378(16)36308-6. No abstract available. PMID 13736585
- [Background] Roberts CL, Algert CS, Nippita TA, Bowen JR, Shand AW. Association of prelabor cesarean delivery with reduced mortality in twins born near term. Obstet Gynecol. 2015 Jan;125(1):103-110. doi: 10.1097/AOG.0000000000000578. PMID 25560111
- [Background] Silver RM. Delivery after previous cesarean: long-term maternal outcomes. Semin Perinatol. 2010 Aug;34(4):258-66. doi: 10.1053/j.semperi.2010.03.006. PMID 20654776
- [Background] Thurmond AS, Harvey WJ, Smith SA. Cesarean section scar as a cause of abnormal vaginal bleeding: diagnosis by sonohysterography. J Ultrasound Med. 1999 Jan;18(1):13-6; quiz 17-8. doi: 10.7863/jum.1999.18.1.13. PMID 9952074
- [Background] van der Voet LF, Bij de Vaate AM, Veersema S, Brolmann HA, Huirne JA. Long-term complications of caesarean section. The niche in the scar: a prospective cohort study on niche prevalence and its relation to abnormal uterine bleeding. BJOG. 2014 Jan;121(2):236-44. doi: 10.1111/1471-0528.12542. PMID 24373597
- [Background] Weiniger CF, Lyell DJ, Tsen LC, Butwick AJ, Shachar B, Callaghan WM, Creanga AA, Bateman BT. Maternal outcomes of term breech presentation delivery: impact of successful external cephalic version in a nationwide sample of delivery admissions in the United States. BMC Pregnancy Childbirth. 2016 Jul 8;16(1):150. doi: 10.1186/s12884-016-0941-9. PMID 27392035